CLINICAL TRIAL: NCT01065259
Title: Randomized Control Study of Concerta and Strattera on the Improvement of Executive Function in Attention Deficit Hyperactivity Disorder Children
Brief Title: Concerta and Strattera on the Executive Function in Attention Deficit Hyperactivity Disorder (ADHD) Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Yufeng Wang, Peking University the Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CON-I-07-CN-029-B
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: attention deficit hyperactivity disorder; executive function; OROS MPH; atomoxetine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OROS MPH (Experimental): the group treated by OROS MPH
  Interventions: Drug: OROS MPH
- atomoxetine (Active Comparator): the group treated by atomoxetine
  Interventions: Drug: Atomoxetine
- control (No Intervention): the normal control with no intervention

INTERVENTIONS:
Drug: OROS MPH — The dosage began with 18mg Qd. It can be increased with 18mg every week until an optimal response achieved. The maximum dosage was no more than 54mg/d. The optimal dosage will maintain for 4 to 6 weeks
  Other Names: Concerta
  Arms: OROS MPH
Drug: Atomoxetine — The dosage begins with 0.5mg/kg.d. It can increased to 0.8mg/kg.d at the second week, 1.2mg/kg.d at the third week, and 1.4mg/kg.d at the 5th week according to the patients response. The optimal dosage will maintain for 4 to 6 weeks.
  Other Names: Strattera
  Arms: atomoxetine

SUMMARY:
The objective of this study is to compare the effect of Concerta (Osmotic Release Oral System Extended Release Methylphenidate HCL, OROS MPH) and Strattera (Atomoxetine) on the laboratory and ecological executive function in children with attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
The sample will include 134 ADHD children and adolescence, randomized assigned to Concerta and strattera treatment group, with 67 cases in each. It will also include 67 sex and age matched normal control. The drug will be titrated to optimal dose. The executive function including inhibition, working memory, set shifting and plan will be compared among two medication group and the control group, using laboratory executive function test and Behavior Rating Inventory of Executive Function (BRIEF).

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 to 16 years old. Body weight between 20 to 60 kg
* Meet ADHD criteria in tne Diagnostic and Statistic Manual of Mental Disorders, fourth edition (DSM-IV) through questionaire and interview
* Intelligence quotient (IQ) >= 70
* Currently unmedicated or effectively medicated with immediately released methylphenidate (The maximum dosage no more than 60mg/d)
* The patient and the parent express their will to comply with the follow up including the clinical interview and all the test
* The parent or the guardian sign the written consent
* Can swallow the capsule

Exclusion Criteria:

* Have administered immediate release methylphenidate, OROS MPH or atomoxetine, but ADHD symptoms not improved.
* Bipolar I or II disorder, psychosis, or pervasive developmental disorder.
* Meet the DSM-IV anxiety disorder.
* Any seizure disorder (except for febrile convulsion) or electroencephalogram (EEG) abnormal associated with epilepsy, or currently taking anti-convulsion drugs.
* Depression disorder, tend to commit suicide, or comorbid depression symptoms which need immediate treatment.
* Tics disorder, or Tourette's syndrom（DSM-IV 307.23）, or family history of tics disorder.
* Narrow-angle glaucoma
* cardiovascular diseases, or any diseases may be deteriorated when the pulse or the blood pressure increased, including hypertension or those taking anti-hypertension drugs.
* Diseases significantly enhance the sympathetic nervous system activity, or taking sympathomimetic drug every day.
* Allergic to methylphenidate or atomoxetine, or serious allergic reaction to more than one drugs or adverse event to multiple drugs before.
* Serious gastrointestinal stenosis
* History of alcohol, drug or other substance abuse
* Those using unprescribed potential abuse drugs in screening.
* In the process of the trial, the patient need to take other psychotropic drug other than the experimental drugs, including health food with central nervous system (CNS) activity (e.g. melatonin).
* Might begin any structure psychological therapy addressed for ADHD in the process of the trial
* Have used other psychotropic drugs in the past 30 days, including monoamine oxidase inhibitor.
* Are participating other clinical trial.
* Have difficulty in following up in 8 weeks.
* Relatives of the investigator.
* Employee of Xi-an Jensen or Eli lilly company.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 262 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Executive function test | seven to ten weeks

SECONDARY OUTCOMES:
ADHD Rating Scale-IV | seven to ten weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yufeng Wang, M.D. PH.D., Principal Investigator — Peking University Institute of Mental Health
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Su Y, Yang L, Stein MA, Cao Q, Wang Y. Osmotic Release Oral System Methylphenidate Versus Atomoxetine for the Treatment of Attention-Deficit/Hyperactivity Disorder in Chinese Youth: 8-Week Comparative Efficacy and 1-Year Follow-Up. J Child Adolesc Psychopharmacol. 2016 May;26(4):362-71. doi: 10.1089/cap.2015.0031. Epub 2016 Jan 18. PMID 26779845
- [Derived] Yang L, Cao Q, Shuai L, Li H, Chan RC, Wang Y. Comparative study of OROS-MPH and atomoxetine on executive function improvement in ADHD: a randomized controlled trial. Int J Neuropsychopharmacol. 2012 Feb;15(1):15-26. doi: 10.1017/S1461145711001490. Epub 2011 Oct 21. PMID 22017969